CLINICAL TRIAL: NCT04849598
Title: Effects of an Automatic Oxygen Titration vs. Constant Oxygen Flow Rates During Daily Activities in Patients After SARS-CoV-2 Infection
Brief Title: Automatic Oxygen Titration in Patients After SARS-CoV-2 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Rembert Koczulla, Head of Pneumological Department, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: O2matic_COVID
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Post-COVID19
Keywords: post SARS-CoV-2 infection; long-term oxygen therapy; automatic oxygen-titration; hypoxemia
MeSH Terms: conditions — Hypoxia | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ESWT Order A and B (Experimental): First Endurance Shuttle Walk Test using the automatic oxygen titration (O2matic) with the target range being 90 - 94% SpO2, the second Endurance Shuttle Walk Test using the prescribed constant flow oxygen therapy.
  Interventions: Other: Oxygen therapy
- ESWT Order B and A (Experimental): First Endurance Shuttle Walk Test using the prescribed constant flow oxygen therapy, the second Endurance Shuttle Walk Test using the automatic oxygen titration (O2matic) with the target range being 90 - 94% SpO2.
  Interventions: Other: Oxygen therapy
- Stairs Order A and B (Experimental): First Stair Walking Test using the automatic oxygen titration (O2matic) with the target range being 90 - 94% SpO2, the second Stair Walking Test using the prescribed constant flow oxygen therapy.
  Interventions: Other: Oxygen therapy
- Stairs Order B and A (Experimental): First Stair Walking Test using the prescribed constant flow oxygen therapy, the second Stair Test using the automatic oxygen titration (O2matic) with the target range being 90 - 94% SpO2.
  Interventions: Other: Oxygen therapy

INTERVENTIONS:
Other: Oxygen therapy — Oxygen therapy during ESWTs and Stair Walking Test: one test using the prescribed constant oxygen flow and one using an automatic oxygen titration system. SpO2 target range: 90 - 94%

SUMMARY:
With the progression of the SARS-CoV-2 pandemic there's an increasing number of patients recovering from COVID19. Some of these patients still experience hypoxemia and therefore are still in need of a long-term oxygen therapy (LTOT), usually provided as a constant-flow. However, during a patient's daily activities, oxygenation levels may vary and the same constant flow may not be suitable for all tasks. Studies in COPD patients suggest that an automatic oxygen titration, which adjusts the oxygen flow automatically according to a patient's blood oxygen levels to prevent desaturations, could be beneficial compared to a constant oxygen titration during exercise.

So far there are no studies available that directly compare the automatic oxygen titration with the patient's prescribed constant oxygen flow in patients with hypoxemia after SARS-CoV-2 infection during activities of daily life. Therefore, the primary outcome of this study is to investigate the effects of an automatic oxygen titration (O2matic, Denmark) in comparison to constant oxygen flow rates as prescribed according to guidelines.

DETAILED DESCRIPTION:
Rationale

After an infection with SARS-CoV-2, some patients still experience hypoxemia even after being discharged from the hospital. Long-term oxygen therapy (LTOT) is then used to increase the patients blood oxygen level and prolong the time spent within the SpO2 target range, decreasing the probability of severe hypoxemia or at least lowering the time spent in this severe hypoxemia and all in all enhance the patient's endurance. A prescription for LTOT is usually given for constant flow rates which might vary during day- and night use.

This study is a randomized, controlled cross-over trial. Its aim is to investigate the effects of an automatic oxygen titration in patients after SARS-CoV-2 infection on the blood oxygen saturation level during activities of daily life (walking). Secondary, the effects of using an automatic titration on endurance, pCO2 blood level as well as heart rate and breathing frequency are compared to using the prescribed constant flow oxygen therapy.

Design:

Each patient undergoes a series of shuttle walk tests. After an initial incremental shuttle walk test (ISWT) to determine the patient's maximum walking speed, the patient undergoes 2 endurance shuttle walk tests (ESWTs) at 85% of the maximum walking speed. One of these ESWTs is performed with the prescribed constant oxygen flow, the other with the O2matic automatic oxygen titration in a random order.

In addition to the shuttle walk tests, patient will perform two stair walking tests, again one with the prescribed constant oxygen flow, the other with the O2matic automatic oxygen titration in a random order.

Furthermore, patients will be asked to rate their experienced comfort after each ESWT and to name their preferred oxygen titration system.

ELIGIBILITY:
Inclusion Criteria:

* validated COVID19 disease in case history
* hypoxemia (PO2 < 55 mmHg) under room air conditions (rest or during exercise) or SpO2 <88% during exercise
* already established Long-term oxygen therapy or given indication for a Long-term oxygen therapy

Exclusion Criteria:

* acute infection
* cardiovascular diseases that limit physical fitness
* orthopedic diseases preventing the patient from undergoing the walking tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Change of oxygen saturation during the endurance shuttle walk Tests | Day 2, 3
  SpO2 measured by continuous transcutaneous recording via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland)

SECONDARY OUTCOMES:
Change of transcutaneous pCO2 during ESWTs | Day 2, 3
  tc pCO2 measured by continuous transcutaneous recording via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland)
Change of heart rate during ESWTs and stair walking tests | Day 2, 3, 4
  Heart rate measured by continuous transcutaneous recording via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland)
Change of respiratory rate during ESWTs | Day 2, 3
  Respiratory rate measured by ApneaLink Air™
Change of time to desaturation (SpO2 ≤ 90%) and to severe desaturation (SpO2 ≤ 85%) during ESWTs and Stair Walking Tests | Day 2, 3, 4
  SpO2 measured by continuous transcutaneous recording via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland) and O2matic Device.
Change of Endurance time (s) | Day 2, 3, 4
  Change of Walking Duration during the ESWT and Stair Walking Tests
Change of capillary partial pressure of CO2 (pCO2) during endurance shuttle walk tests | Day 2, 3
  pCO2 measured by capillary blood gases taken before and after the ESWT
Change of capillary partial pressure of O2 (pO2) during endurance shuttle walk tests | Day 2,3
  pO2 measured by capillary blood gases taken before and after the ESWT
Patients preference due to oxygen delivery system | Day 3
  Patients will be asked to rate their experienced comfort after each ESWT
Change of number of stairs | Day 4
  Change of the number of stairs the patient was able to climb during Stair Walking Tests

CONTACTS AND LOCATIONS:
Overall Officials: Andreas R Koczulla, Prof. Dr. med., Principal Investigator — Philipps University Marburg
Locations (1):
- Klinikum Berchtesgadener Land, Schön Kliniken, Schönau am Königssee, Bavaria, Germany

REFERENCES:
- [Background] Lellouche F, L'Her E, Bouchard PA, Brouillard C, Maltais F. Automatic Oxygen Titration During Walking in Subjects With COPD: A Randomized Crossover Controlled Study. Respir Care. 2016 Nov;61(11):1456-1464. doi: 10.4187/respcare.04406. Epub 2016 Oct 18. PMID 27794080
- [Background] Singh SJ, Puhan MA, Andrianopoulos V, Hernandes NA, Mitchell KE, Hill CJ, Lee AL, Camillo CA, Troosters T, Spruit MA, Carlin BW, Wanger J, Pepin V, Saey D, Pitta F, Kaminsky DA, McCormack MC, MacIntyre N, Culver BH, Sciurba FC, Revill SM, Delafosse V, Holland AE. An official systematic review of the European Respiratory Society/American Thoracic Society: measurement properties of field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1447-78. doi: 10.1183/09031936.00150414. Epub 2014 Oct 30. PMID 25359356
- [Background] Prieur G, Combret Y, Medrinal C, Arnol N, Bonnevie T, Gravier FE, Quieffin J, Lamia B, Reychler G, Borel JC. Energy conservation technique improves dyspnoea when patients with severe COPD climb stairs: a randomised crossover study. Thorax. 2020 Jun;75(6):510-512. doi: 10.1136/thoraxjnl-2019-214295. Epub 2020 Mar 26. PMID 32217783